CLINICAL TRIAL: NCT02476474
Title: Antral Length and GERD Following Sleeve Gastrectomy for Morbid
Brief Title: GERD Following Laparoscopic Sleeve Gastrectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn due to a lack of funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 133508
Record Dates: First submitted 2015-06-03; First posted 2015-06-19 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 cm start of resection (Active Comparator): The line of resection for the Laparoscopic Sleeve gastrectomy will start at 3 cm from pylorus (antrum).
  Interventions: Procedure: 3 cm start of resection
- 6 cm start of resection (Active Comparator): The line of resection for the Laparoscopic Sleeve gastrectomy will start at 6 cm from pylorus (antrum).
  Interventions: Procedure: 6 cm start of resection

INTERVENTIONS:
Procedure: 3 cm start of resection — Investigators will start the resection of the LSG 3 centimeters from the antrum of the stomach.
  Arms: 3 cm start of resection
Procedure: 6 cm start of resection — Investigators will start the resection of the LSG 6 centimeters from the antrum of the stomach.
  Arms: 6 cm start of resection

SUMMARY:
Laparoscopic Sleeve Gastrectomy (LSG) creates a vertical gastrectomy which results in a narrow and tubular shape of stomach. The line of resection starts at 3-6 cm. from pylorus (antrum) toward to the angle of His. The gastric antrum plays a major role in gastric emptying, particularly for solids. Hence, depending upon the starting point of gastric sleeve resection in each center, this can result in difference of the remaining gastric antrum which may affect gastric emptying time after this procedure.

DETAILED DESCRIPTION:
Laparoscopic Sleeve Gastrectomy (LSG), a purely restrictive procedure, has become recently one of the most popular bariatric surgical procedures in this decade because its surgical technique is simple but outcomes in regards to weight loss and co-morbidities improvement are excellent comparable to other procedures. Nevertheless, this procedure carries one potential drawback namely "gastroesophageal reflux disease (GERD). The impact on GERD following LSG are inconsistent . Additionally, the recent literature can be divided into two categories: those that support an increase in GERD prevalence after LSG and those that demonstrate a decrease in GERD prevalence after LSG. Postoperatively, one of the proposed mechanisms for either increased or decreased GERD prevalence is gastric emptying time. Delayed gastric emptying time can contribute to increase intra-gastric volume and pressure resulting in an increase in prevalence of GERD after surgery. On the other hand, accelerated gastric emptying time can cause decrease in GERD prevalence because of decrease in stomach volume and interorgan pressure after operation. In addition, LSG creates a vertical gastrectomy which results in a narrow and tubular shape of stomach. The line of resection starts at 3-6 cm. from pylorus (antrum) toward to the angle of His. The gastric antrum plays a major role in gastric emptying, particularly for solids. Hence, depending upon the starting point of gastric sleeve resection in each center, this can result in difference of the remaining gastric antrum which may affect gastric emptying time after this procedure. The investigators hypothesize that a larger amount of gastric antrum will result in accelerated gastric emptying time which leads to less GERD prevalence. On the contrary, the less the remaining gastric antrum would result in delayed gastric emptying which contribute to more GERD prevalence. The investigators plan on identifying the prevalence of GERD in the patients who undergo LSG comparing those who have the sleeve beginning either 3 cm. or 6 cm. from pylorus. We will utilize 24 hour esophageal pH monitoring, esophageal manometry, upper gastrointestinal scintigraphy and esophagogastroduodenoscopy at preoperatively, 3 and 6 month postoperatively. Ultimately, this study will help further clarify the most proper starting resected point of LSG (3 versus 6 cm. from pylorus) which results in the least GERD prevalence after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any subject who has already been already cleared for and scheduled to undergo laparoscopic sleeve gastrectomy for the treatment of morbid obesity(Utilizing NIH1991 guideline for bariatric surgery)

Exclusion Criteria:

1. Patients not meeting entry criteria to undergo bariatric surgery procedures.
2. Refusal to give informed consent.
3. Age <18 or >70.
4. Prior small intestinal or gastric resective surgery
5. Existing coagulopathy (INR>2.0, platelet count<100,000)
6. Severe reflux esophagitis.( Los Angeles Classification for erosive esophagitis grade C,D)
7. Hiatal hernia > 2 cm(according to esophageal manometry or EGD)
8. Acquired or Congenital Immunodeficiencies
9. White blood cell count below normal range.
10. Azotemia - serum creatinine > 2.0 mg/dl

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time of gastric emptying | 6 months post surgery

SECONDARY OUTCOMES:
Number of participants with GERD | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John P Cello, MD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Background] Melissas J, Daskalakis M, Koukouraki S, Askoxylakis I, Metaxari M, Dimitriadis E, Stathaki M, Papadakis JA. Sleeve gastrectomy-a "food limiting" operation. Obes Surg. 2008 Oct;18(10):1251-6. doi: 10.1007/s11695-008-9634-4. Epub 2008 Jul 29. PMID 18663545
- [Background] Laffin M, Chau J, Gill RS, Birch DW, Karmali S. Sleeve gastrectomy and gastroesophageal reflux disease. J Obes. 2013;2013:741097. doi: 10.1155/2013/741097. Epub 2013 Jul 15. PMID 23956846
- [Background] Chiu S, Birch DW, Shi X, Sharma AM, Karmali S. Effect of sleeve gastrectomy on gastroesophageal reflux disease: a systematic review. Surg Obes Relat Dis. 2011 Jul-Aug;7(4):510-5. doi: 10.1016/j.soard.2010.09.011. Epub 2010 Sep 21. PMID 21130052
- [Background] Braghetto I, Davanzo C, Korn O, Csendes A, Valladares H, Herrera E, Gonzalez P, Papapietro K. Scintigraphic evaluation of gastric emptying in obese patients submitted to sleeve gastrectomy compared to normal subjects. Obes Surg. 2009 Nov;19(11):1515-21. doi: 10.1007/s11695-009-9954-z. Epub 2009 Aug 28. PMID 19714384
- [Background] Weiner RA, Weiner S, Pomhoff I, Jacobi C, Makarewicz W, Weigand G. Laparoscopic sleeve gastrectomy--influence of sleeve size and resected gastric volume. Obes Surg. 2007 Oct;17(10):1297-305. doi: 10.1007/s11695-007-9232-x. PMID 18098398
- [Background] Bernstine H, Tzioni-Yehoshua R, Groshar D, Beglaibter N, Shikora S, Rosenthal RJ, Rubin M. Gastric emptying is not affected by sleeve gastrectomy--scintigraphic evaluation of gastric emptying after sleeve gastrectomy without removal of the gastric antrum. Obes Surg. 2009 Mar;19(3):293-8. doi: 10.1007/s11695-008-9791-5. Epub 2008 Dec 17. PMID 19089519